CLINICAL TRIAL: NCT03309618
Title: Improving Arterial Wall Characteristics in Patients After Myocardial Infarction With a Very Low Dose of Fluvastatin and Valsartan: Proof-of-concept Study
Brief Title: Post- Myocardial Infarction Arterial Wall Improvement by Low-dose Fluvastatin and Valsartan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Martina Turk Veselič, Principal Investigator, M.D., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGE-MI
Record Dates: First submitted 2017-10-04; First posted 2017-10-13 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; arterial stiffness; pulse wave velocity; flow mediated dilatation; fluvastatin; valsartan
MeSH Terms: conditions — Myocardial Infarction | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treatment group (Experimental): 20 participants received low-dose combination of fluvastatin (10 mg) and valsartan (20 mg) (low-flu/val) per orally once daily for 30 days.
  Interventions: Drug: low-dose combination of fluvastatin (10 mg) and valsartan (20 mg) (low-flu/val)
- Control group (Placebo Comparator): 16 participants received placebo per orally once daily for 30 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: low-dose combination of fluvastatin (10 mg) and valsartan (20 mg) (low-flu/val)
  Arms: Treatment group
Drug: placebo
  Arms: Control group

SUMMARY:
The concept of improving arterial wall characteristics by treatment with a very low-dose combination of fluvastatin and valsartan (low-flu/val) in stable, post-myocardial infarction (MI) patients was tested. The parameters of endothelial function (flow mediated dilatation (FMD), reactive hyperemia index) and arterial stiffness (carotid-femoral pulse wave velocity (cf-PWV), local carotid PWV and β-stiffness coefficient) were measured before and after 30 days of treatment, and the residual effect was assessed 10 weeks later. So the investigators explored whether low-flu/val added "on-top-of" optimal therapy could improve endothelial function and arterial stiffness in post-MI patients. Since these improved parameters are well-known predictors of future coronary events, such treatment could decrease cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* history of MI in the last 0.5 to 5 years
* males
* aged under 55 years

Exclusion Criteria:

* diabetes mellitus
* manifest peripheral artery disease or carotid artery disease
* acute infection
* chronic diseases
* present therapy with fluvastatin and/or valsartan.

Max Age: 55 Years | Sex: Male
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
brachial flow mediated dilatation (FMD) | 30 days
  ultrasonographically measured flow mediated dilatation of brachial artery
carotid pulse wave velocity (c-PWV) | 30 days
  ultrasonographically measured pulse wave velocity of carotid artery
β-stiffness coefficient | 30 days
  ultrasonographically measured β-stiffness coefficient of carotid artery
carotid-femoral pulse wave velocity (cf-PWV) | 30 days
  carotid-femoral pulse wave velocity measured by Sphygmocor
reactive hyperemia index (RHI) | 30 days
  reactive hyperemia index measured by an Endopat device

SECONDARY OUTCOMES:
brachial flow mediated dilatation (FMD) | 10 weeks after termination of intervention
  ultrasonographically measured flow mediated dilatation of brachial artery
carotid pulse wave velocity (c-PWV) | 10 weeks after termination of intervention
  ultrasonographically measured pulse wave velocity of carotid artery
β-stiffness coefficient | 10 weeks after termination of intervention
  ultrasonographically measured β-stiffness coefficient of carotid artery
carotid-femoral pulse wave velocity (cf-PWV) | 10 weeks after termination of intervention
  carotid-femoral pulse wave velocity measured by Sphygmocor
reactive hyperemia index (RHI) | 10 weeks after termination of intervention
  reactive hyperemia index measured by an Endopat device

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vascular Diseases, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neunteufl T, Heher S, Katzenschlager R, Wolfl G, Kostner K, Maurer G, Weidinger F. Late prognostic value of flow-mediated dilation in the brachial artery of patients with chest pain. Am J Cardiol. 2000 Jul 15;86(2):207-10. doi: 10.1016/s0002-9149(00)00857-2. No abstract available. PMID 10913483
- [Background] Bonetti PO, Lerman LO, Lerman A. Endothelial dysfunction: a marker of atherosclerotic risk. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):168-75. doi: 10.1161/01.atv.0000051384.43104.fc. PMID 12588755
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] Stefanadis C, Dernellis J, Tsiamis E, Stratos C, Diamantopoulos L, Michaelides A, Toutouzas P. Aortic stiffness as a risk factor for recurrent acute coronary events in patients with ischaemic heart disease. Eur Heart J. 2000 Mar;21(5):390-6. doi: 10.1053/euhj.1999.1756. PMID 10666353
- [Background] Orlova IA, Nuraliev EY, Yarovaya EB, Ageev FT. Prognostic value of changes in arterial stiffness in men with coronary artery disease. Vasc Health Risk Manag. 2010 Nov 4;6:1015-21. doi: 10.2147/VHRM.S13591. PMID 21127698
- [Background] Li Z, Iwai M, Wu L, Liu HW, Chen R, Jinno T, Suzuki J, Tsuda M, Gao XY, Okumura M, Cui TX, Horiuchi M. Fluvastatin enhances the inhibitory effects of a selective AT1 receptor blocker, valsartan, on atherosclerosis. Hypertension. 2004 Nov;44(5):758-63. doi: 10.1161/01.HYP.0000145179.44166.0f. Epub 2004 Sep 27. PMID 15452025
- [Background] Inaba Y, Chen JA, Bergmann SR. Prediction of future cardiovascular outcomes by flow-mediated vasodilatation of brachial artery: a meta-analysis. Int J Cardiovasc Imaging. 2010 Aug;26(6):631-40. doi: 10.1007/s10554-010-9616-1. Epub 2010 Mar 26. PMID 20339920
- [Background] Lunder M, Janic M, Savic V, Janez A, Kanc K, Sabovic M. Very low-dose fluvastatin-valsartan combination decreases parameters of inflammation and oxidative stress in patients with type 1 diabetes mellitus. Diabetes Res Clin Pract. 2017 May;127:181-186. doi: 10.1016/j.diabres.2017.03.019. Epub 2017 Mar 22. PMID 28384560
- [Background] Lunder M, Janic M, Jug B, Sabovic M. The effects of low-dose fluvastatin and valsartan combination on arterial function: a randomized clinical trial. Eur J Intern Med. 2012 Apr;23(3):261-6. doi: 10.1016/j.ejim.2011.11.011. Epub 2011 Dec 12. PMID 22385885
- [Background] Boncelj Svetek M, Erzen B, Kanc K, Sabovic M. Impaired endothelial function and arterial stiffness in patients with type 2 diabetes - The effect of a very low-dose combination of fluvastatin and valsartan. J Diabetes Complications. 2017 Mar;31(3):544-550. doi: 10.1016/j.jdiacomp.2016.12.002. Epub 2016 Dec 16. PMID 28012835
- [Background] Janic M, Lunder M, Cerkovnik P, Prosenc Zmrzljak U, Novakovic S, Sabovic M. Low-Dose Fluvastatin and Valsartan Rejuvenate the Arterial Wall Through Telomerase Activity Increase in Middle-Aged Men. Rejuvenation Res. 2016 Apr;19(2):115-9. doi: 10.1089/rej.2015.1722. Epub 2016 Jan 22. PMID 26214555